CLINICAL TRIAL: NCT04483180
Title: Sweeteners and Sweetness Enhancers: Short-term Impact on Food Behaviour, Physiology & Health (Phase 1)
Brief Title: Work Package 2 Phase 1 - Beverages Study
Acronym: SWEET-WP2-P1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Leeds (Other); University of Copenhagen (Other); University of Liverpool (Other); University of Surrey (Other); Bioiatriki HEALTHCARE GROUP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 774293-WP2-P1
Record Dates: First submitted 2020-07-08; First posted 2020-07-23 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2020-06

CONDITIONS: Glycemic Index; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Cross-Over Studies

STUDY DESIGN:
Intervention Model Description: Multi-centre crossover study with 4 conditions using balanced block randomisation. The three centres will follow different randomisation sequences but will all test the same 4 conditions (University of Navarra, University of Copenhagen, University of Liverpool).
Who Masked: Participant, Investigator
Masking Description: Double blind study. Neither the participant nor the investigator will be aware of the coding of beverages used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Beverage containing a sucrose solution. Same aspect and flavor than the experimental beverages. About 1/4 of participants will start with this beverage first.
  Interventions: Other: Comparison of sweetener blends in liquid form (cross-over study)
- Sucralose / acesulfame K (Experimental): Beverage containing a blend of sweeteners based on sucralose and acesulfame K. Same aspect and flavour than the control beverage. About 1/4 of participants will start with this beverage first.
  Interventions: Other: Comparison of sweetener blends in liquid form (cross-over study)
- Stevia rebaudioside A / thaumatin (Experimental): Beverage containing a blend of sweeteners based on stevia rebaudioside A and thaumatin. Same aspect and flavour than the control beverage. About 1/4 of participants will start with this beverage first.
  Interventions: Other: Comparison of sweetener blends in liquid form (cross-over study)
- Mogroside V / stevia rebaudioside M (Experimental): Beverage containing a blend of sweeteners based on mogroside V and stevia rebaudioside M. Same aspect and flavour than the control beverage. About 1/4 of participants will start with this beverage first.
  Interventions: Other: Comparison of sweetener blends in liquid form (cross-over study)

INTERVENTIONS:
Other: Comparison of sweetener blends in liquid form (cross-over study) — The aim is to compare the effects of different sweetener blends on glycemia, subjective appetite parameters and safety parameters when consumed in a beverage as part of a breakfast

SUMMARY:
Within the SWEET project (EU funded), in Work Package 2 there are two phases, this study refers to Phase 1 of the SWEET WP2 project, which will be a coordinated trial across 3 intervention centres, University of Navarra (UNAV), University of Liverpool (ULIV) and University of Copenhagen (UCPH). It will involve an acute intervention in 120 individuals to explore initial acceptance, safety and post-prandial effects of 3 S&SE blends delivered in beverage format.

The main endpoints of the SWEET WP2 Phase 1 study will be glycaemic and lipaemic responses; eating behavior (subjective appetite, food preference, cravings, reward), and health effects (rebound hunger, G.I. side effects and metabolic effects). This phase will be exploratory and will not involve any specific primary hypotheses.

DETAILED DESCRIPTION:
This protocol has the overall objective to evaluate the acute (short-term, 1 day) and repeated (medium-term, 2 week) effects of combinations of sweeteners and sweetness enhancers (S&SEs) on metabolic, sensory and neuro-behavioural processes involved in satiety, consumer preference and health, and to explore mechanistic processes, genetic background, safety issues and consumer perspectives.

There are 4 products being tested in 4 different formulations (sucrose-sweetened beverage control vs. 3 reformulated beverages with S&SE). Each product will be tested at 3 intervention sites in double-blind cross-over trials with 40 subjects per site, tested per product. Therefore a total of 120 subjects will take part across the 3 intervention sites (UNAV, ULIV, UCPH).

Using identical procedures each trial will consist of 4 Clinical Investigation Days (CIDs) scheduled 7-11 days apart for each of the 3 product formulations.

The total duration of WP2 Phase 2 per site is 6 months, including a minimum of 22 days and a maximum of 34 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years.
* BMI: 25 to 35 kg/m2.
* For women: Use of contraceptive methods or not planning to become pregnant for the duration of the study.
* Regular consumption of sugar-containing foods and willing to consume artificially-sweetened beverages (a score of ≥ 5 on the short sFFQ Part 1a and answer Yes to all questions in Part 2).
* Able to participate on the visit days/CIDs during normal working hours.
* Healthy as determined from the self-reported medical history or when a clinical condition exists, when this is considered to be irrelevant (i.e. not influencing study outcomes) for the study by the study medical doctor.
* Consuming breakfast regularly (at least 5 days per week).
* Liking of the study foods defined by a response of Yes for each of the breakfast foods during the pre-screening interview and a score of 40 % or above on the Liking VAS for the control beverage.
* Able to understand and be willing to sign the informed consent form, and to follow all the study procedures and requirements.

Exclusion Criteria:

* Blood donation < 3 month prior to study.
* Deficient nutrition or hydration status as identified from the pre-screening/screening session (i.e. absence of disease including anaemia, BMI >18 kg/m2, or other criteria as determined by the study doctor).
* Food allergy, intolerance, restriction or avoidance of any of the study foods (e.g. veganism) or history of anaphylactic reaction to any food.
* Likelihood for disordered eating defined as a score of 20 or more on the EAT-26 test.
* Currently dieting to lose weight or having been on weight cycles (i.e. repeatedly lost and re-gained weight) in the last 3 months.
* Smoking.
* Binge drinking i.e. consuming >14 units of alcohol per week in women or >21 units/week in men less than 4 days apart.
* Performing >10 h of intense physical activity per week.
* Continuous night or late shift work (ending later than 11 pm on a permanent basis). Rotational shift work allowed if can attend on days that do not follow a late/night shift.
* Self-reported use of drugs of abuse within the previous 12 months.
* For women: Pregnancy, lactation.
* Persons who do not have access to either (mobile) phone or internet (this is necessary when being contacted by the study personnel during the study).
* Insufficient communication in the national language.
* Proven or suspected inability, physically or mentally, to comply with the procedures required by the study protocol as evaluated by the daily study manager, site-PI, PI or clinical responsible. This includes volunteers for which insufficient collaboration may be foreseen.
* Subject's general condition contraindicates continuing in the study as evaluated by the daily study manager, site-PI, PI or clinical responsible.
* Simultaneous participation in other relevant clinical intervention studies.
* Previous university or college training related to eating behaviour research.
* Medical conditions as known by the person:

  * Self-reported eating disorders.
  * Diagnosed anaemia.
  * Diagnosed diabetes mellitus.
  * Abnormal gastro-intestinal (G.I) function or structure such as malformation, angiodysplasia, active peptic ulcer.
  * Active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption.
  * History of G.I. surgery with permanent effect (i.e. surgical treatment of obesity).
  * Medical history of cardio-vascular disease (e.g. current angina; myocardial infarction or stroke within the past 6 months; heart failure; symptomatic peripheral vascular disease).
  * Significant liver disease, e.g. cirrhosis (fatty liver disease allowed).
  * Malignancy which is currently active or in remission for less than five years after last treatment (local basal and squamous cell skin cancer allowed).
  * Thyroid diseases, except those on Levothyroxine treatment of hypothyroidism if the person has been on a stable dose for at least 3 months.
  * Psychiatric illness (e.g. major depression, bipolar disorders).
* Medication:

  * Use currently or within the previous 3 months of prescription or over the counter medication that has the potential of affecting appetite, satiety or body weight incl. food supplements.

Except: low dose antidepressants if they, in the judgement of the daily study manager, site-PI, PI or clinical responsible, do not affect weight or following the study protocol. Levothyroxine for treatment of hypothyroidism is allowed if the person has been on a stable dose for at least 3 months.

• Cholesterol lowering medication, if the dose has changed during the last 3 months (i.e. the medication is allowed if the participant has been on a stable dose for at least 3 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose area under the curve (AUC) | Clinical Investigation Day 1, 2, 3, 4
  Area Under the Curve (AUC) for blood glucose (120 min post-intake)
Blood Insulin AUC | Clinical Investigation Day 1, 2, 3, 4
  Area Under the Curve for blood Insulin (120 min post-intake)
Hunger iAUC | Clinical Investigation Day 1, 2, 3, 4
  Incremental Area Under the Curve for hunger (120 min post-intake)
Fasting Blood glucose | Clinical Investigation Day 1, 2, 3, 4
  Fasting blood glucose
30 min Blood glucose | Clinical Investigation Day 1, 2, 3, 4
  Blood glucose at 30 min post-intake
60 min Blood glucose | Clinical Investigation Day 1, 2, 3, 4
  Blood glucose at 60 min post-intake
90 min Blood glucose | Clinical Investigation Day 1, 2, 3, 4
  Blood glucose at 90 min post-intake
120 min Blood glucose | Clinical Investigation Day 1, 2, 3, 4
  Blood glucose at 120 min post-intake
Fasting Blood insulin | Clinical Investigation Day 1, 2, 3, 4
  Fasting blood insulin
30 min Blood insulin | Clinical Investigation Day 1, 2, 3, 4
  Blood insulin at 30 min post-intake
60 min Blood insulin | Clinical Investigation Day 1, 2, 3, 4
  Blood insulin at 60 min post-intake
90 min Blood insulin | Clinical Investigation Day 1, 2, 3, 4
  Blood insulin at 90 min post-intake
120 min Blood insulin | Clinical Investigation Day 1, 2, 3, 4
  Blood insulin at 120 min post-intake
Fasting Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Fasting subjective appetite questionnaire. Visual Analogue Scale
5 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 5 min post-intake
15 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 15 min post-intake
30 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 30 min post-intake
45 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 45 min post-intake
60 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 60 min post-intake
120 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 120 min post-intake
180 min Hunger (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Subjective appetite questionnaire. Visual Analogue Scale at 180 min post-intake

SECONDARY OUTCOMES:
Fasting Blood cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Fasting blood cholesterol
30 min Blood cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Blood cholesterol at 30 min post-intake
60 min Blood cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Blood cholesterol at 60 min post-intake
90 min Blood cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Blood cholesterol at 90 min post-intake
120 min Blood cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Blood cholesterol at 120 min post-intake
Fasting Triglycerides | Clinical Investigation Day 1, 2, 3, 4
  Fasting triglycerides in serum
30 min Triglycerides | Clinical Investigation Day 1, 2, 3, 4
  Triglycerides in serum at 30 min post-intake
60 min Triglycerides | Clinical Investigation Day 1, 2, 3, 4
  Triglycerides in serum at 60 min post-intake
90 min Triglycerides | Clinical Investigation Day 1, 2, 3, 4
  Triglycerides in serum at 90 min post-intake
120 min Triglycerides | Clinical Investigation Day 1, 2, 3, 4
  Triglycerides in serum at 120 in post-intake
Fasting HDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Fasting HDL-cholesterol in serum
30 min HDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  HDL-cholesterol in serum at 30 min post-intake
60 min HDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  HDL-cholesterol in serum at 60 min post-intake
90 min HDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  HDL-cholesterol in serum at 90 min post-intake
120 min HDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  HDL-cholesterol in serum at 120 min post-intake
Fasting LDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  Fasting LDL-cholesterol in serum
30 min LDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  LDL-cholesterol in serum at 30 min post-intake
60 min LDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  LDL-cholesterol in serum at 60 min post-intake
90 min LDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  LDL-cholesterol in serum at 90 min post-intake
120 min LDL-cholesterol | Clinical Investigation Day 1, 2, 3, 4
  LDL-cholesterol in serum at 120 min post-intake
Fasting Alanine aminotransferase (ALT) | Clinical Investigation Day 1, 2, 3, 4
  Fasting liver function marker ALT
120 min Alanine aminotransferase (ALT) | Clinical Investigation Day 1, 2, 3, 4
  Liver function marker ALT at 120 min post-intake
Fasting Aspartate aminotransferase (AST) | Clinical Investigation Day 1, 2, 3, 4
  Fasting liver function marker AST
120 min Aspartate aminotransferase (AST) | Clinical Investigation Day 1, 2, 3, 4
  Liver function marker AST at 120 min post-intake
Weight | Visit 0 (screening), Clinical Investigation Day 4
  Anthropometry marker
Height | Visit 0 (screening)
  Anthropometry marker
Body Mass Index (BMI) | Visit 0 (screening), Clinical Investigation Day 4
  Anthropometry marker
Waist Circumference (WC) | Visit 0 (screening)
  Anthropometry marker
Hip Circumference (HC) | Visit 0 (screening)
  Anthropometry marker
Waist-to-hip ratio (WHR) | Visit 0 (screening)
  Anthropometry marker
Leeds Food Preference Questionnaire (LFPQ) | Clinical Investigation Day 1, 2, 3, 4
  Change in food preference and food reward at 15-20 min post-intake
Liking (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Liking and explicit wanting of the beverage at 5 min post-intake
Fasting FG21 | Clinical Investigation Day 1, 2, 3, 4
  Fasting FG21 concentration in serum
30 min FG21 | Clinical Investigation Day 1, 2, 3, 4
  FG21 concentration in serum at 30 min post-intake
60 min FG21 | Clinical Investigation Day 1, 2, 3, 4
  FG21 concentration in serum at 60 min post-intake
90 min FG21 | Clinical Investigation Day 1, 2, 3, 4
  FG21 concentration in serum at 90 min post-intake
120 min FG21 | Clinical Investigation Day 1, 2, 3, 4
  FG21 concentration in serum at 120 min post-intake

OTHER OUTCOMES:
Consumers' Perspectives Questionnaire | Visit 0 (screening)
  Psychological health drivers (perceptions)
Blood DNA Analysis | Clinical Investigation Day 1
  DNA analysis for genetic polymorphism presence
24 hour food recall | Next day after each clinical investigation day (1, 2, 3, 4)
  Interview to know what the volunteers ate during the 24h following the beverage intake
24 hour Gastro Intestinal side effects | Next day after each clinical investigation day (1, 2, 3, 4)
  Interview to know if the volunteers experienced side effects during the 24h following the beverage intake
End of day questionnaire (VAS registered) | Clinical Investigation Day 1, 2, 3, 4
  Food cravings during the 8 h following the beverage intake
Risk factors for chronic disease | Visit 0 (screening)
  Baseline weight, height, BMI, WC and WHR, physical activity
Socio-demographic questionnaire | Visit 0 (screening)
  Ethnicity, household and employment
Eating Attitudes Test-26 (EAT-26) | Visit 0 (screening)
  Eating behaviour traits
Short sugar Food Frequency Questionnaire (short sFFQ) | Visit 0 (screening)
  Habitual intake of sweet foods
End of study survey | Clinical Investigation Day 4
  Perception and evaluation of the clinical trial
Taste test (VAS registered) | Visit 0 (screening)
  Liking of the study beverage

CONTACTS AND LOCATIONS:
Locations (3):
- University of Copenhagen, Frederiksberg, Denmark
- Centre for Nutrition Research, University of Navarra, Pamplona, Navarre, Spain
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Almiron-Roig E, Navas-Carretero S, Castelnuovo G, Kjolbaek L, Romo-Hualde A, Normand M, Maloney N, Hardman CA, Hodgkins CE, Moshoyiannis H, Finlayson G, Scott C, Raats MM, Harrold JA, Raben A, Halford JCG, Martinez JA. Impact of acute consumption of beverages containing plant-based or alternative sweetener blends on postprandial appetite, food intake, metabolism, and gastro-intestinal symptoms: Results of the SWEET beverages trial. Appetite. 2023 May 1;184:106515. doi: 10.1016/j.appet.2023.106515. Epub 2023 Feb 26. PMID 36849009